CLINICAL TRIAL: NCT01874210
Title: Study on Colonic Fermentation in Chronic Kidney Disease Patients
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S51367
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Fecal sample, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hemodialysis: Hemodialysis patients
- Control: 1. Household contacts on the same diet
  2. Healthy unrelated controls

SUMMARY:
Chronic kidney disease is associated with the accumulation of various metabolites, i.e., uremic retention solutes. Evidence is mounting that the colonic microbiome contributes substantially to these uremic retention solutes. Indoxyl sulfate and p-cresyl sulfate are among the most extensively studied gut microbial metabolites, and are associated with cardiovascular disease, chronic kidney disease progression and overall mortality. Indirect findings suggest that chronic kidney disease influences the colonic microbial metabolism with higher p-cresyl sulfate urinary excretion rates at more advanced renal disease. Therefore, this study aims to elucidate the influence of renal dysfunction on microbial metabolism and to test the hypothesis that chronic kidney disease patients carry a different fecal metabolite profile.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 95 years
* Treatment with renal replacement therapy, i.e. hemo- or peritoneal dialysis for more than 3 months
* Written informed consent

Exclusion Criteria:

* History of organic gastro-intestinal disease (e.g., inflammatory bowel disease, malignancy)
* History of colonic surgery
* Recipient of a renal or other solid organ transplant
* Use of pre-/pro-/syn- or antibiotics in preceding 4 weeks

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients treated with renal replacement therapy, i.e. hemo- or peritoneal dialysis for more than 3 months
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2008-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
difference in fecal metabolite profile (Chronic kidney disease vs. control) | baseline
  difference in fecal metabolite profile between chronic kidney disease patients and control group

SECONDARY OUTCOMES:
difference in fecal metabolite profile depending on dialysis modality | baseline
  difference in fecal metabolite profile between hemodialysis patients and peritoneal patients

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Poesen, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Björn Meijers, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Kristin Verbeke, Pharm PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Pieter Evenepoel, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium